CLINICAL TRIAL: NCT01857232
Title: Randomised, Double-blind, Dose-finding Phase II Study to Assess the Efficacy of APD403 in the Prevention of Nausea and Vomiting Caused by Cisplatin- or Anthracycline/Cyclophosphamide (AC)-Based Chemotherapy
Brief Title: Dose-finding Study of APD403 to Prevent Nausea and Vomiting After Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DN10016
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: CINV
MeSH Terms: interventions — Ondansetron; Dexamethasone; fosaprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (Other): OND + DEX + FOS followed by oral DEX
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Fosaprepitant
- Placebo (Placebo Comparator): OND + APD403 followed by oral PLACEBO
  Interventions: Drug: Ondansetron; Drug: Placebo; Drug: APD403 IV
- Low dose APD403 (Experimental): OND + APD403 followed by oral APD403 low dose
  Interventions: Drug: Ondansetron; Drug: APD403 IV; Drug: APD403 oral
- Mid dose APD403 (Experimental): OND + APD403 followed by oral APD403 mid dose
  Interventions: Drug: Ondansetron; Drug: APD403 IV; Drug: APD403 oral
- High dose APD403 (Experimental): OND + APD403 followed by oral APD403 high dose
  Interventions: Drug: Ondansetron; Drug: APD403 IV; Drug: APD403 oral

INTERVENTIONS:
Drug: Ondansetron — 5HT3-antagonist
Drug: Placebo — Comparator
  Arms: Placebo
Drug: Dexamethasone — Corticosteroid
  Arms: Control
Drug: Fosaprepitant — NK1 antagonist
  Arms: Control
Drug: APD403 IV — Amisulpride IV 20 mg
  Arms: High dose APD403; Low dose APD403; Mid dose APD403; Placebo
Drug: APD403 oral — Amisulpride oral 10, 20 or 40 mg
  Arms: High dose APD403; Low dose APD403; Mid dose APD403

SUMMARY:
Comparison of efficacy of APD403 at preventing delayed sickness in patients who have received cancer chemotherapy

ELIGIBILITY:
Inclusion criteria

* Male or female patients ≥ 18 years of age
* Ability and willingness to give written informed consent
* Patients scheduled to receive, on day 1 of their chemotherapy, either: (i) a first cisplatin chemotherapy infusion at a dose of ≥70 mg/m2 (males and females); or (ii) a first infusion of cyclophosphamide at a dose of 500-1500 mg/m2 in combination with either epirubicin at a dose of 60-100 mg/m2 or doxorubicin at a dose of 40-60 mg/m2 (females only)
* Karnofsky performance score ≥ 60%
* Adequate cardiac, hepatic and renal function

  * QTc interval < 500 ms
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) < 5 x upper limit normal (ULN)
  * Bilirubin < 5 x ULN
  * Creatinine < 3 x ULN
* Adequate haematological function

  * Haemoglobin ≥ 8 g/dL
  * White blood count ≥ 3.0 x 109/L
  * Platelet count ≥ 100 x 109/L
* For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner) or a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom) during the study and for a period of at least 48 hours afterwards

Exclusion Criteria

* Patients scheduled to receive, prior to or in the 120 hours after cisplatin or AC, any other chemotherapeutic agent with a high or moderate emetic risk
* Patients who have previously received anti-neoplastic chemotherapy
* Patients scheduled to receive paclitaxel or docetaxel during the first cycle of their chemotherapy
* Patients undergoing abdominal or pelvic irradiation within 48 hours prior to screening or scheduled to receive abdominal or pelvic irradiation between screening and 24 hours after cisplatin or AC administration
* Patients with a known prolactin-dependent tumour (e.g. pituitary gland prolactinoma or confirmed prolactin-dependent breast cancer) or phaeochromocytoma
* Patients with a pre-existing vestibular disorder
* Patients being treated with regular anti-emetic therapy including corticosteroids
* Patients receiving inhaled corticosteroids, unless started more than one month prior to the expected date of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Herrstedt, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Herrstedt J, Summers Y, Jordan K, von Pawel J, Jakobsen AH, Ewertz M, Chan S, Naik JD, Karthaus M, Dubey S, Davis R, Fox GM. Amisulpride prevents nausea and vomiting associated with highly emetogenic chemotherapy: a randomised, double-blind, placebo-controlled, dose-ranging trial. Support Care Cancer. 2019 Jul;27(7):2699-2705. doi: 10.1007/s00520-018-4564-8. Epub 2018 Nov 28. PMID 30488222

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: ACUTE (day 1): IV OND + FOS + DEX
  • DELAYED (days 2 to 4): Oral DEX
- Placebo: ACUTE (day 1): IV OND + APD403 20 mg DELAYED (days 2 to 4): Oral Placebo
- APD403 10MG: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral APD403 10 mg
- APD403 20MG: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral APD403 20 mg
- ADP403 40MG: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral APD403 40 mg
Period: Overall Study
Arm/Group | Control | Placebo | APD403 10MG | APD403 20MG | ADP403 40MG
Started | 69 | 67 | 67 | 70 | 69
Evaluable ITT | 66 | 66 | 63 | 68 | 65
Completed | 61 | 65 | 63 | 68 | 63
Not Completed | 8 | 2 | 4 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control ( Dexamethazon): ACUTE (day 1): IV OND + FOS + DEX
  • DELAYED (days 2 to 4): Oral DEX
- Total: Total of all reporting groups
Arm/Group | Control ( Dexamethazon) | Placebo | APD403 10MG | APD403 20MG | ADP403 40MG | Total
Number analyzed (Participants) | 66 | 66 | 63 | 68 | 65 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (10.38) | 57.3 (11.01) | 56.9 (11.24) | 56.6 (10.53) | 56.5 (10.59) | 57.1 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 52 | 52 | 51 | 257
  Male | 15 | 15 | 11 | 16 | 14 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 65 | 64 | 62 | 68 | 64 | 323
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: Participants]
  Denmark | 16 | 12 | 13 | 17 | 15 | 73
  Germany | 23 | 23 | 19 | 21 | 22 | 108
  United Kingdom | 27 | 31 | 31 | 30 | 28 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delayed Phase Complete Response(CR)
Description: Delayed phase complete response (CR), defined as an absence of emetic episodes and no rescue medication use in the period from 24 to 120 hours after the initiation of chemotherapy.
  The primary endpoint was analysed separately in the strata of chemotherapy regimen and gender, and in the strata of country.
Time Frame: 24-120 hours
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- PLACEBO: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral Placebo
- ADP421 20MG: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral APD403 20 mg
- APD421 40MG: ACUTE (day 1): IV OND + APD403 20 mg
  • DELAYED (days 2 to 4): Oral APD403 40 mg
Arm/Group | Control | PLACEBO | APD403 10MG | ADP421 20MG | APD421 40MG
Number analyzed (Participants) | 66 | 66 | 63 | 68 | 65
Participants | 37 | 13 | 27 | 21 | 20
Statistical Analysis 1: Comparison: PLACEBO vs APD403 10MG; Test type: Superiority; p = 0.004, Regression, Logistic
Statistical Analysis 2: Comparison: PLACEBO vs ADP421 20MG; Test type: Superiority; p = 0.0987, Regression, Logistic
Statistical Analysis 3: Comparison: PLACEBO vs APD421 40MG; Test type: Superiority; p = 0.1041, Regression, Logistic

2. Secondary Outcome: Number of Participants With CR in the Overall Phase.
Description: CR defined as no emesis and no use of rescue medication, in the overall phase (0 to 120 hours after the initiation of chemotherapy)
Time Frame: 0 to 120 hours after the initiation of chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Placebo | APD403 10MG | APD403 20MG | ADP403 40MG
Number analyzed (Participants) | 66 | 66 | 63 | 68 | 65
Participants | 33 | 11 | 21 | 17 | 17
Statistical Analysis 1: Comparison: Placebo vs APD403 10MG; Test type: Superiority; p = 0.0235, Chi-squared, Corrected; 1-sided
Statistical Analysis 2: Comparison: Placebo vs APD403 20MG; Test type: Superiority; p = 0.1651, Chi-squared, Corrected; 1-sided
Statistical Analysis 3: Comparison: Placebo vs ADP403 40MG; Test type: Superiority; p = 0.1332, Chi-squared, Corrected; 1-sided

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Control | Placebo | APD403 10MG | APD403 20MG | ADP403 40MG
All-Cause Mortality (participants affected / at risk) | 2/66 | 0/66 | 0/63 | 0/68 | 0/65
Serious Adverse Events (participants affected / at risk) | 8/66 | 12/66 | 2/63 | 3/68 | 4/65
Other Adverse Events (participants affected / at risk) | 36/66 | 47/66 | 34/63 | 21/68 | 28/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=66) | Placebo (N=66) | APD403 10MG (N=63) | APD403 20MG (N=68) | ADP403 40MG (N=65)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatine Increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Prolactin Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General Physical Condition Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=66) | Placebo (N=66) | APD403 10MG (N=63) | APD403 20MG (N=68) | ADP403 40MG (N=65)
Fatigue (General disorders) | 13 (13) | 13 (13) | 13 (13) | 5 (5) | 11 (11)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5) | 7 (7) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (7) | 3 (3) | 2 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Mucosal Dryness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 9 (9) | 7 (7) | 3 (3) | 8 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
There were no limitations and caveats with this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days